CLINICAL TRIAL: NCT05114122
Title: Clinical Outcomes of Premolars Restored With Ceramic Vonlay Restorations Versus Onlay Using Modified USPHS Criteria (Randomized Clinical Trial)
Brief Title: Clinical Outcomes of Premolars Restored With Ceramic Vonlay Restorations Versus Onlay Using Modified USPHS Criteria
Acronym: vonlay-onlay
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Abdel Aziz Hazzaa, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-27-10-2020
Record Dates: First submitted 2021-10-27; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Clinical Performance of Ceramic Vonlays
Keywords: Ceramics, vonlay, onlay, fracture
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vonlay lithium disilicate ceramic restorations (Experimental): Vonlay is a hybrid of an onlay with an extended buccal veneer surface for use in bicuspid regions where there is mostly enamel to bond to. The vonlay is less invasive, more readily repairable, less technique-sensitive to attain adequate bonding, and will leave sounder tooth structure remaining if further treatment is required in the future
  Interventions: Procedure: Vonlay Ceramic restorations
- Onlay lithium disilicate ceramic restorations (Active Comparator): Onlays are used to restore large areas of decay and also used to replace old restorations, whether they are defective amalgam fillings, old cast-gold onlays, or fabricated from some other material
  Interventions: Procedure: Onlay Ceramic restorations

INTERVENTIONS:
Procedure: Vonlay Ceramic restorations — vonlay is a hybrid of an onlay with an extended buccal veneer surface for use in bicuspid regions where there is mostly enamel to bond to. The vonlay is less invasive, more readily repairable, less technique-sensitive to attain adequate bonding, and will leave sounder tooth structure remaining if further treatment is required in the future
  Other Names: Onlay ceramic restorations with buccal veneer
  Arms: Vonlay lithium disilicate ceramic restorations
Procedure: Onlay Ceramic restorations — Onlays are used to restore large areas of decay and also used to replace old restorations, whether they are defective amalgam fillings, old cast-gold onlays, or fabricated from some other material
  Arms: Onlay lithium disilicate ceramic restorations

SUMMARY:
Evaluation the clinical performance of premolars restored with ceramic vonlays versus onlays using modified USPHS criteria after follow-up period of 0,3,6,9,12 months

DETAILED DESCRIPTION:
two groups of patients with vital premolars indicated for fixed restorations will be selected according to special inclusion criteria (n=13) in each group (total of 26). one group will receive minimally invasive cavity preparations for posterior indirect restorations either vonlay or onlay according to each group the patient will be assessed using Modified USPHS Criteria at 0,3,6,9,12 months regarding fracture, marginal integrity and marginal discoloration

ELIGIBILITY:
Inclusion Criteria:

1. Age range of the patients from 25-44 years old, who could read understand and write to sign the consent by himself /herself
2. Have no active periodontal or pulpal diseases, have teeth with good restorations.(19)
3. Psychologically and physically able to withstand conventional dental procedures
4. Patients with teeth problems indicated for onlay and vonlay (premolars).

   1. Decayed teeth.
   2. Teeth restored with large filling restorations.
5. Able to return for follow-up examinations and evaluation.

Exclusion Criteria:

1. Patient less than 25 or more than 44 years.
2. Patient with active resistant periodontal diseases.
3. Patients with poor oral hygiene, high caries risk and uncooperative patients.
4. Pregnant women.
5. Patients in the growth stage with partially erupted teeth.
6. Psychiatric problems or unrealistic expectations.
7. Lack of opposing dentition in the area of interest. 8- The presence of a removable or fixed orthodontic appliance, signs of bruxism or clenching, the absence of more than one unit in the posterior region

Ages: 25 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Fracture | change from baseline at 3,6,9,12 months
  assessed according to modified USPHS criteria (Alpha, Bravo)

SECONDARY OUTCOMES:
Marginal integrity | 0,3,6,9,12 months
  assessed according to modified USPHS criteria (Alpha, Bravo, Charlie and Delta)
Marginal discoloration | 0,3,6,9,12 months
  assessed according to modified USPHS criteria (Alpha, Bravo and Charlie)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, 11 El-Saraya St. El Manial, Cairo, El Manial, Egypt